CLINICAL TRIAL: NCT05307874
Title: A Two-part, Open-label, Clinical Study to Assess the Safety, Tolerability and Activity of Intravenous Doses of ICT01 in Combination With Low-dose Subcutaneous Interleukin-2 in Patients With Advanced Solid Tumors (EVICTION-2)
Brief Title: Phase 1/2a Study of ICT01 Plus Low Dose SC IL-2 in Patients With Advanced Solid Tumors
Acronym: EVICTION-2
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ImCheck Therapeutics (Industry)
Collaborators: ILife Consulting (Unknown); Exystat (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ICT01-102
Record Dates: First submitted 2022-03-24; First posted 2022-04-01 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumor, Adult
MeSH Terms: interventions — Interleukin-2; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- Dose level 2 ICT01 + Low dose SC IL-2 (Experimental): For all arms, ICT01 IV is given on Day 1 of every 21-day cycle. SC IL-2 is administered Days 1-5 of cycles 1/2/3 only.
  Interventions: Drug: ICT01; Drug: Proleukin Injectable Product
- Dose Level 1 ICT01 + High dose SC IL-2 (Experimental): For all arms, ICT01 IV is given on Day 1 of every 21-day cycle. SC IL-2 is administered Days 1-5 of cycles 1/2/3 only.
  Interventions: Drug: ICT01; Drug: Proleukin Injectable Product
- Dose level 1 ICT01 + Low dose SC IL-2 (Experimental): For all arms, ICT01 IV is given on Day 1 of every 21-day cycle. SC IL-2 is administered Days 1-5 of cycles 1/2/3 only.
  Interventions: Drug: ICT01; Drug: Proleukin Injectable Product
- Dose level 3 ICT01 + Low dose SC IL-2 (Experimental): For all arms, ICT01 IV is given on Day 1 of every 21-day cycle. SC IL-2 is administered Days 1-5 of cycles 1/2/3 only.
  Interventions: Drug: ICT01; Drug: Proleukin Injectable Product
- Dose level 4 ICT01 + Low dose SC IL-2 (Experimental): For all arms, ICT01 IV is given on Day 1 of every 21-day cycle. SC IL-2 is administered Days 1-5 of cycles 1/2/3 only.
  Interventions: Drug: ICT01; Drug: Proleukin Injectable Product
- Dose level 5 ICT01 + Low dose SC IL-2 (Experimental): For all arms, ICT01 IV is given on Day 1 of every 21-day cycle. SC IL-2 is administered Days 1-5 of cycles 1/2/3 only.
  Interventions: Drug: ICT01; Drug: Proleukin Injectable Product
- Primer Dose level 2 ICT01+ Low dose SC IL-2 + Booster Dose level 2 ICT01 (Experimental): ICT01 IV is given on Day 1 of every 21-day cycle and on day 8 of Cycles 1-3. SC IL-2 is administered on Days 1-5 of Cycles 1/2/3 only.
  Interventions: Drug: ICT01; Drug: Proleukin Injectable Product
- Primer Dose level 2 ICT01+ Low dose SC IL-2 + Booster Dose level 3 ICT01 (Experimental): ICT01 IV is given on Day 1 of every 21-day cycle and on day 8 of Cycles 1-3. SC IL-2 is administered on Days 1-5 of Cycles 1/2/3 only.
  Interventions: Drug: ICT01; Drug: Proleukin Injectable Product
- Dose level 2 ICT01 + Low dose SC IL-2 + Pembrolizumab (Experimental): ICT01 IV and Pembrolizumab are given on Day 1 of every 21-day cycle. SC IL-2 is administred Days 1-5 of cycles 1/2/3 only.
  Interventions: Drug: ICT01; Drug: Proleukin Injectable Product; Drug: Pembrolizumab injection
- Dose level 4 ICT01 + Low dose SC IL-2 + Pembrolizumab (Experimental): ICT01 IV and Pembrolizumab are given on Day 1 of every 21-day cycle. SC IL-2 is administred Days 1-5 of cycles 1/2/3 only.
  Interventions: Drug: ICT01; Drug: Proleukin Injectable Product; Drug: Pembrolizumab injection
- Primer Dose level 2 ICT01+ Low dose SC IL-2 + Pembrolizumab + Booster Dose level 2 ICT01 (Experimental): ICT01 IV and Pembrolizumab are given on Day 1 of every 21-day cycle. ICT01 IV is given on day 8 of Cycles 1-3. SC IL-2 is administered on Days 1-5 of Cycles 1/2/3 only.
  Interventions: Drug: ICT01; Drug: Proleukin Injectable Product; Drug: Pembrolizumab injection

INTERVENTIONS:
Drug: ICT01 — anti-BTN3A mAb IV Q3W
Drug: Proleukin Injectable Product — 1 MIU/m2 SC IL-2 daily x 5 days for the first 3 cycles
  Other Names: IL-2
Drug: Pembrolizumab injection — 200mg administered following ICT01 + LDSC IL-2 over 30 min Q3W
  Arms: Dose level 2 ICT01 + Low dose SC IL-2 + Pembrolizumab; Dose level 4 ICT01 + Low dose SC IL-2 + Pembrolizumab; Primer Dose level 2 ICT01+ Low dose SC IL-2 + Pembrolizumab + Booster Dose level 2 ICT01

SUMMARY:
This is a phase I/IIa, two-part, open-label study to characterize the safety, tolerability, pharmacodynamics, and antitumor activity of ICT01 in combination with LDSC IL-2 in patients with advanced-stage solid tumors.

Part 1 will be a dose escalation of IV ICT01 administered on the first day of every 21-day cycle (CnD1) to patients with advanced-stage solid tumors in combination with LDSC IL-2 (Proleukin®) administered daily on days 1-5 of cycles 1-3 (C1-3D1-5). Objectives of part 1 are to characterize the safety of the combination regimen and determine the RP2D for Part 2.

Part 2 will comprise a maximum of 2 indications and 2 combination dosing regimens of ICT01 +LDSC IL-2, which will be supported by statistical power calculations once the indications are selected. The final regimen will be ICT01 + LDSC IL-2 + Pembrolizumab on a Q3W cycle. The primary objective of Part 2 is to demonstrate the efficacy of the combination regimen based on RECIST1.1 in one or more solid tumor indications.

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed/refractory patients who have failed at least 2 lines of systemic therapy or who failed first line therapy and are intolerant of or have a contraindication to the standard second line of therapy with histologically or cytologically confirmed diagnosis of:

   1. metastatic colorectal cancer (CRC):
   2. metastatic ovarian cancer:
   3. metastatic castration-resistant prostate cancer (mCRPC)
   4. metastatic pancreatic ductal adenocarcinoma (PDAC)
   5. metastatic or unresectable refractory melanoma

      2) Availability of baseline tumor biopsy and willingness to undergo on-study tumor biopsies 3) Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1 4) Life expectancy > 3 months as assessed by the Investigator 5) At least 1 measurable lesion per RECIST1.1

      Exclusion Criteria:
      1. Any malignancy of γ9δ2 T cell origin
      2. Any systemic anti-tumor-directed drug therapy within 28 days or 5 times the elimination half-life (whichever is shorter) before study treatment
      3. Treatment with investigational drugs within 28 days before study treatment
      4. Systemic steroids at a daily dose of > 10 mg of prednisone, > 2 mg of dexamethasone or equivalent, for the last 28 days and ongoing
      5. Patients with rapidly progressing disease defined as advanced/metastatic, symptomatic, visceral spread, with a risk of life-threatening complications in the short term (e.g., during Screening Period/ treatment washout) that includes patients with massive uncontrolled effusions pleural, pericardial, peritoneal, pulmonary lymphangitis, and over 50% liver involvement
      6. Ongoing immune-related adverse events (irAEs) ≥grade 2 not resolved from previous therapies except vitiligo, stable neuropathy up to grade 2, hair loss, and stable endocrinopathies with substitutive hormone therapy.
      7. Ongoing systemic autoimmune disease requiring systemic immunosuppressive therapy
      8. Primary or secondary immune deficiency
      9. Active and uncontrolled infections requiring intravenous antibiotic or antiviral treatment
      10. Patients with contraindication to IL-2 treatment according to the SmPC/package insert

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2022-05-04 (Actual); Primary Completion 2025-10-09 (Actual); Study Completion 2025-10-09 (Actual)

PRIMARY OUTCOMES:
Treatment-Emergent Adverse Events | 1 year
  Incidence and severity of adverse events related to study treatment

SECONDARY OUTCOMES:
Change from baseline in the number of circulating g9d2 T cells | Cycle Days 8 & 15 for the first 3 cycles
  flow cytometry measurement of circulating and intratumoral g9d2 T cells
Disease Control Rate | 1 year
  Stable disease or better by RECIST1.1

CONTACTS AND LOCATIONS:
Overall Officials: Katrien Lemmens, MD, PhD, Study Director — ImCheck Therapeutics
Locations (5):
- France (2):
  - Institute Gustave Roussy, Paris
  - IUCT Oncopole Claudius Regaud, Toulouse
- Germany (2):
  - University Carl Gustav Carus, Dresden
  - Universitätsklinikum Wuerzburg, Würzburg
- The Institute of Cancer Research, Sutton, United Kingdom

REFERENCES:
- [Background] De Gassart A, Le KS, Brune P, Agaugue S, Sims J, Goubard A, Castellano R, Joalland N, Scotet E, Collette Y, Valentin E, Ghigo C, Pasero C, Colazet M, Guillen J, Cano CE, Marabelle A, De Bonno J, Hoet R, Truneh A, Olive D, Frohna P. Development of ICT01, a first-in-class, anti-BTN3A antibody for activating Vgamma9Vdelta2 T cell-mediated antitumor immune response. Sci Transl Med. 2021 Oct 20;13(616):eabj0835. doi: 10.1126/scitranslmed.abj0835. Epub 2021 Oct 20. PMID 34669444